CLINICAL TRIAL: NCT03936972
Title: In the Cost-conscious Era: Ilizarov Circular Frame or Uniplanar External Fixator for Management of Open Tibia Shaft Fracture, Retrospective Cohort Study From a Level-1 Trauma Center
Brief Title: Ilizarov Frame or Uni Planar External Fixator in the Cost-conscious Era
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Obada Hasan, FCPS, MRCS, Senior Resident, Aga Khan University
Other Study IDs: 5120 29-Dec-17
Record Dates: First submitted 2019-05-02; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Tibia Fracture
Keywords: tibia fracture; ilizarov; open fracture; external fixator
MeSH Terms: conditions — Tibial Fractures; Fractures, Open

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ilizarov circular frame: 46 participants with open tibia fracture Gustillo type III only
  Interventions: Procedure: ilizarov circular frame and uni-planarexternal fixator
- Ex. Fix: 47 participants with open tibia fracture Gustillo type III only
  Interventions: Procedure: ilizarov circular frame and uni-planarexternal fixator

INTERVENTIONS:
Procedure: ilizarov circular frame and uni-planarexternal fixator — both are types of external fixators, but one is circular frame and other is uni-planar frame

SUMMARY:
Tibial shaft fracture is a common injury worldwide. Their treatment, prognosis, and outcome are determined by the mechanism of injury, presence of communition, soft tissue injury and displacement. In developing countries, lack of education,socioeconomic backgrounds, delay in presentation and appropriate planning for surgery add further to complicate the situation and may end in delayed union, non-union, multiple surgeries and ultimate results in increased morbidity. This study was conducted to determine the outcome of open tibia shaft fracture treated with Ilizarov or AO External Fixator.

DETAILED DESCRIPTION:
Tibial shaft fracture is a common injury worldwide. Their treatment, prognosis, and outcome are determined by the mechanism of injury, presence of communition, soft tissue injury and displacement. In developing countries, lack of education,socioeconomic backgrounds, delay in presentation and appropriate planning for surgery add further to complicate the situation and may end in delayed union, non-union, multiple surgeries and ultimate results in increased morbidity. This study was conducted to determine the outcome of open tibia shaft fracture treated with Ilizarov or AO External Fixator. It was retrospective Cohort study. Two groups were compared in terms of fracture healing, mechanism of injury, fracture classification, Participant's ambulation at discharge, New Injury Severity Score (NISS), duration of hospital stay, duration of fracture union, need for secondary procedures and complications. Investigators concluded that circular fixator application has favorable outcomes for Gustilo grade III open tibial shaft fractures as compared to uniplanar external fixator.

ELIGIBILITY:
Inclusion Criteria:

Participants with open tibia shaft fracture type III (A, B, C) as per Gustillo classification of open fractures stabilized with external fixation either circular or uniplanar external fixator were included

Exclusion Criteria:

* All closed and type I and II open tibia shaft fractures according to Gustillo classification of open fracture, Intra-articular fracture extending to knee and ankle joints were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult participants both genders presenting with open fracture of tibia specifically Gustillo type III (Severe injury).
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
fracture healing | 6-9 months
  Radiographic union score (RUST) for tibial fractures was used. months later on non-union.

SECONDARY OUTCOMES:
Union | 6-9 months
  Union was defined fracture healing after 6 months and delayed union after 9

IPD SHARING:
Plan to Share IPD: No
Not allowed as per hospital policy